CLINICAL TRIAL: NCT03139565
Title: A Randomized Controlled Trial Comparing High-dose vs. Standard Influenza Vaccine in Adult Solid Organ Transplant Recipients
Brief Title: High Dose vs. Standard Influenza Vaccine in Adult SOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Deepali Kumar, Physician, Transplant Infectious Diseases, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UHNTID004
Record Dates: First submitted 2017-04-06; First posted 2017-05-04 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Influenza; Immunosuppression
Keywords: Influenza; Solid Organ Transplant; Infection; Vaccine; Immunogenicity
MeSH Terms: conditions — Influenza, Human; Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluzone High-dose Influenza Vaccine (Experimental): This treatment consists of 60 microgram of each influenza antigen provided as a single injection, which will be injected in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Fluzone High-dose Influenza Vaccine
- Standard 2016-2017 Flu vaccine (Active Comparator): This will be the Standard 2016-2017 influenza vaccine made available by public health. It will contain 15 microgram of each strain and will be delivered in the deltoid muscle of non-dominant arm.
  Interventions: Biological: Standard 2016-2017 Flu vaccine

INTERVENTIONS:
Biological: Fluzone High-dose Influenza Vaccine — This treatment consists of 60 microgram of each influenza antigen provided as a single injection, which will be injected in the deltoid muscle of the non-dominant arm.
  Arms: Fluzone High-dose Influenza Vaccine
Biological: Standard 2016-2017 Flu vaccine — The intramuscular preparation of the vaccine used for the control group will be the Standard influenza vaccine made available by public health. The intramuscular dose (standard 0.5 mL) will contain 15 microgram antigen from each strain and delivered in the deltoid muscle by trained personnel.
  Arms: Standard 2016-2017 Flu vaccine

SUMMARY:
The study will test whether a high dose influenza vaccination results in improved immunogenicity in adult SOT recipients as compared to standard vaccine. This will be a single center prospective observer-blind randomized controlled trial conducted at the Toronto General Hospital Multi-Organ Transplant Unit, University Health Network, Toronto, Ontario, Canada.

DETAILED DESCRIPTION:
Influenza virus is an important cause of morbidity and mortality in the transplant population and can lead to viral and bacterial pneumonia. Although the annual influenza vaccine is recommended for transplant patients, studies have shown that standard vaccine has poor immunogenicity. Currently, there are no studies that define the effect of high-dose vaccine in adult transplant recipients even though this population could potentially benefit from it. The study will compare the immunogenicity of two different types of the influenza vaccine in 240 solid organ transplant patients during the 2016-2017 season. Patients will be randomized to receive either high-dose or standard dose influenza vaccine. Antibody titers will be evaluated by a standard hemagglutination inhibition assay. The hypothesis is that the patients who receive the high-dose influenza vaccine will reach a significantly greater response to the vaccine. This study advances research on the prevention of serious viral infections in transplant recipients. Results from this study have the potential to directly improve patient care. If the use of the high-dose influenza vaccine is successful, this strategy may lead to significant reduction in burden of disease, hospitalization, and long-term morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Organ transplant recipient on at least one immunosuppressive
* Age >=18
* Outpatient status
* Greater than 3 months post transplant

Exclusion Criteria:

* Has already received influenza vaccination for 2016-2017 season
* Egg allergy or allergy to previous influenza vaccine
* Febrile illness in the past one week
* Active Cytomegalovirus viremia
* Use of Rituximab in the past 6 months
* Ongoing or recent (in past 30 days) therapy for acute rejection
* Chronic kidney insufficiency (creatinine clearance ≤30mL/min or dialysis-dependent
* Previous life-threatening reaction to influenza vaccine (i.e. Guillain Barre Syndrome)
* Receipt of intravenous immunoglobulin (IVIG) in the past 30 days or planning to receive IVIG in the next 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Vaccine Immunogenicity (antibody titers) | 4 weeks
  Comparing pre-vaccine and 4 weeks Post-Vaccine antibody titers. Positive vaccine response will be defined as:
  * Seroconversion rate of 4-fold or greater increase in HAI antibody titers to each of the three antigens in the vaccine, and
  * seroprotection rate determined by HAI tigers of 1>=40 post immunization

SECONDARY OUTCOMES:
Vaccine Safety (local and systemic adverse events to vaccination). | 6 months
  Vaccine Safety assessed by local and systemic adverse events to vaccination.
Vaccine Safety (rates of rejection). | 6 months
  Vaccine Safety assessed by rates of biopsy proven allograft rejection in the 6 months following vaccination.
Vaccine Immunogenicity (CMI) | 4 weeks
  Analysis of cell-mediated immunity (CMI) in subgroup of 50 patients at 4 weeks post-vaccination vs pre-vaccination samples. CMI response will be correlated with HAI response.
Vaccine Efficacy (influenza infection) | 6 months
  Microbiology proven influenza infection in the 6 months following vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto General Hospital, Multi-Organ Transplant, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natori Y, Shiotsuka M, Slomovic J, Hoschler K, Ferreira V, Ashton P, Rotstein C, Lilly L, Schiff J, Singer L, Humar A, Kumar D. A Double-Blind, Randomized Trial of High-Dose vs Standard-Dose Influenza Vaccine in Adult Solid-Organ Transplant Recipients. Clin Infect Dis. 2018 May 17;66(11):1698-1704. doi: 10.1093/cid/cix1082. PMID 29253089